CLINICAL TRIAL: NCT02896504
Title: Chemotherapy Effect on Brain Structure, Neurophysiology and Psychomotor Behavior in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: R-739-12
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Chemobrain; Chemotherapy; Hormonal Therapy; Neuroimaging
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Chemotherapy: Breast Cancer patients undergoing conventional postsurgical adjuvant chemotherapy treatment
  Interventions: Drug: Exposure: Adjuvant chemotherapy treatment
- Hormonal Therapy: Breast Cancer patients undergoing conventional postsurgical adjuvant hormonal therapy treatment (with no Chemotherapy)
  Interventions: Drug: Exposure: Adjuvant hormonal therapy treatment
- Healthy Control: Healthy age, height and body-mass matched healthy controls

INTERVENTIONS:
Drug: Exposure: Adjuvant chemotherapy treatment
  Groups: Chemotherapy
Drug: Exposure: Adjuvant hormonal therapy treatment
  Groups: Hormonal Therapy

SUMMARY:
Some cancer patients report experiencing mild problems with thinking during or following chemotherapy. Symptoms include problems concentrating, slow thinking, some gaps in memory and difficulty performing complex or multi-tasks. These symptoms often soon disappear after treatment. However for some patients, they may persist for years and this can have a significant effect on their quality of life. The reasons for these symptoms are not well understood.

This study proposes to examine the effects of chemotherapy on the brain and how the changes in the brain affect one's ability to move one's arms and fingers. By better understanding the negative consequences of chemotherapy on the brain and nervous system, the hope is to help pharmaceutical companies develop safer cancer treatment drugs.

DETAILED DESCRIPTION:
Adjuvant chemotherapy (CTh) is an established postoperative treatment often prescribed to cancer patients to reduce risk of relapse. However, a great proportion of patients report experiencing cognitive, psychomotor, and other functional impairments associated with CTh. Some symptoms may persist for years after treatment and can have dramatic consequences on cancer survivors' quality of life. Despite numerous studies reporting various symptoms during/after CTh treatment, mechanisms underlying these symptoms are not well understood. Recent animal and human brain imaging studies suggest that CTh may have direct neurotoxic effects on the brain, in particular on brain white matter (WM). However, to date, no longitudinal studies have been done to examine the effects of CTh on cortical/subcortical WM integrity in human patients. Furthermore, no effort has yet been made to correlate a given WM structure with its corresponding neurophysiological function (NPF) and behavior. This study proposes longitudinal experiments in women diagnosed with breast cancer to examine the effects of CTh on the corpus callosum (CC) and corticospinal tract (CST) (Aim 1), on NPF that directly depends on the quality of CC/CST structure, and on psychomotor behavior critically relying on CC/CST function (conductivity) (Aim 2). The relationship between CC/CST structural integrity and their corresponding NPF and psychomotor behavior will also be examined (Aim 3). The general underlying hypotheses of the study are that (1) CTh has a direct neurotoxic effect on the CC and CST, resulting in microstructural degeneration and (2) structural damage to the CC and CST impairs relevant neurophysiological function and behavior. This research is expected to yield significant information regarding neural structural and physiological causes of CTh-related side effects; known this information would help more effectively manage the symptoms. By demonstrating direct evidence of detrimental consequences of CTh on the central nervous system, it is hoped that the evidence would encourage pharmaceutical companies to develop safer cancer treatment drugs.

ELIGIBILITY:
Inclusion Criteria:

* For all participants

  1. Female aged 20-70
  2. Right handed as determined by the Edinburgh Inventory [40]
  3. Proficient in English
* For Cancer patients

  1. Had breast cancer surgery
  2. Stage I, II, IIIa
  3. Non metastatic cancer
  4. Chemotherapy Patients: Scheduled to receive or receiving breast cancer chemotherapy with Anthracycline and/or Taxane
  5. Hormonal Therapy Patients: Scheduled to receive or receiving hormonal therapy with Aromatase inhibitor
  6. For patients recruited before adjuvant therapy: Adjuvant therapy starts at least 2 weeks after surgery
  7. For patients recruited after adjuvant therapy started: Before completing/within 1 month post chemotherapy Within 4 months after starting hormonal therapy

Exclusion Criteria:

1. Symptoms for mild or severe depression as determined by a Patient Health Questionnaire (PHQ-8) score >14
2. Significant impairment in ability to understand and analyze information as determined by a Folstein Mini-Mental State Exam score <21.
3. Prior history of cancer (except breast cancer for breast cancer patients), trauma, neurological, psychiatric, physical or psychological diseases or other conditions that may influence nervous system structure and function
4. Current medication believed to affect cognitive/psychomotor function (i.e., opioid analgesics, anxiolytics or antidepressants)
5. History of alcohol, smoking and drug abuse
6. Transcranial Magnetic Stimulation or MRI contraindication

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Change in Structural Integrity of the Corpus Collusum as measure by MRI-DTI | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)
Change in Structural Integrity of the cortico-spinal tract as measure by MRI-DTI | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)
Change in out-of-phase bimanual finger tapping task performance | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)
Change in interhemispheric EEG coherence between the left and right motor brain areas | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)
Change in corticomuscular conduction time using Transcranial Magnetic Stimulation | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)
Change in response time to a simple reaction time | Pre to Post chemotherapy change (or at 6 months for hormonal therapy/control)

CONTACTS AND LOCATIONS:
Overall Officials: Guang Yue, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided